CLINICAL TRIAL: NCT04996056
Title: An Open-Label, Randomized Pilot Study Comparing the Safety of a Single Dose of TNX-1300 to Usual Care (UC) Alone for the Treatment of Signs and Symptoms of Acute Cocaine Intoxication in Male Emergency Department (ED) Subjects
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not able to recruit qualified participants
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNX-CE-CI201
Record Dates: First submitted 2021-08-03; First posted 2021-08-09 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Cocaine Intoxication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TNX-1300 (Experimental): TNX-1300 Intravenous injection 200 mg once over 2 mins
  Interventions: Drug: TNX-1300
- Usual Care (Other): Usual Care per the Emergency Department protocol for treating Cocaine Intoxication
  Interventions: Other: Usual Care

INTERVENTIONS:
Drug: TNX-1300 — TNX 1300 200 mg Intravenous injection
  Arms: TNX-1300
Other: Usual Care — Usual Care per the Emergency Department protocol for Cocaine Intoxication
  Arms: Usual Care

SUMMARY:
An Open-Label, Randomized Pilot Study Comparing the Safety of a Single Dose of TNX-1300 to Usual Care (UC) Alone for the Treatment of Signs and Symptoms of Acute Cocaine Intoxication in Male Emergency Department (ED) Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male (sex assigned at birth).
2. Subject is 18-50 years of age.
3. Subject has the capacity to provide voluntary written informed consent.
4. At Screening, subject presents with a SIS total score of ≥6 and a score >1 on at least 1 of the 3 cardiovascular items (HR, systolic and diastolic BP).
5. At Screening, subject presents with cardiac symptoms not present prior to cocaine intoxication, with or without behavioral symptoms.
6. Subject has a positive urine drug screen test at Screening to confirm cocaine use and detect polysubstance abuse (subject may test positive for cannabinoids or opiates).
7. Subject is a suitable candidate for investigational treatment based on the opinion of the investigator.

Exclusion Criteria:

1. Subject who has been admitted to the ED involuntarily.
2. Subject who participated in this clinical study previously.
3. Subject received naloxone (Narcan) within 3 hours prior to informed consent.
4. Subject tests positive for 3,4-Methylenedioxymethamphetamine (MDMA) or amphetamine at Screening.
5. Subject has a prior or current clinically significant untreated cardiac condition. Untreated hypertension may be allowed if not considered severe or life threatening.
6. Subject incurred or is likely to incur a myocardial infarction or other life-threatening severe event or has acute ECG changes indicative of acute coronary syndrome according to investigator judgment.
7. Subject has a clinically significant or unstable medical illness, condition, or disorder that would be anticipated to potentially compromise subject safety or adversely affect the evaluation of clinical outcome parameters.
8. Subject requires physical restraints due to physiological and/or behavioral symptoms.
9. Participation in another investigational drug study (current or within 30 days of Screening).

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events, Adverse Events of Special Interests, and Adverse Drug Reactions | Baseline to 12 Hours
  Incidence of Treatment Emergent Adverse Events, Adverse Events of Special Interests, and Adverse Drug Reactions

SECONDARY OUTCOMES:
Reduction of cardiovascular and other signs and symptoms associated with acute cocaine intoxication identified at Baseline on the Stimulant Intoxication Scale (SIS) | Baseline to 6 Hours
  Reduction of cardiovascular and other signs and symptoms associated with acute cocaine intoxication identified at Baseline on the Stimulant Intoxication Scale (SIS)
Reduction of circulating cocaine, cocaethylene, and EME levels after 15, 60, 120, 240, and 360 minutes in the TNX-1300 arm compared to Baseline | Baseline to 6 Hours
  Reduction of circulating cocaine, cocaethylene, and EME levels after 15, 60, 120, 240, and 360 minutes in the TNX-1300 arm compared to Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sullivan, MD, Study Director — Medical Monitor
Locations (2):
- United States (2):
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri